CLINICAL TRIAL: NCT06653933
Title: Study of Sleep Quality in the Intensive Care Unit and Association with Weaning from Invasive Ventilation in Patients with Chronic Obstructive Bronchopneumopathy.
Acronym: SLEECOP
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: EssaiClinique_SLEECOP
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: COPD; COPD Exacerbation; Ventilated Patients; Ventilator-Associated Pneumonia (VAP); Ventilator Weaning; Weaning of Mechanical Ventilation; Sleep Quality; Sleep Disorders, Circadian Rhythm; Sleep Disorders; Failure, Respiratory; ICU Hospitalization; ICU Sedation
Keywords: COPD; Sleep Quality; Weaning of Mechanical Ventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pneumonia, Ventilator-Associated; Sleep Initiation and Maintenance Disorders; Sleep Disorders, Circadian Rhythm; Sleep Wake Disorders; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- COPD patients with invasive mechanical ventilation in ICU: All patients with COPD who received invasive mechanical ventilation for more than 24 hours in the intensive care unit.

SUMMARY:
Patients admitted in ICU may require invasive mechanical ventilation, using a mechanical ventilator and an endotracheal tube.

In ICU, a prolonged duration of invasive mechanical ventilation may be responsible for ventilator-induced lung injury, pulmonary infection, prolonged administration of sedation, neuromyopathy and prolonged length of stay. The goal of the ICU healthcare teams is therefore to reduce the duration of invasive mechanical ventilation as much as possible.

ICU patients have many sleep disturbances: sleep fragmentation, sleep stage changes, changes in sleep architecture. These sleep disturbances are due to sedation and analgesia, delirium, patient care activities, noise and altered day-night cycles.

Chronic obstructive pulmonary disease (COPD) is a common respiratory disease. COPD complicates the management of invasive mechanical ventilation, particularly weaning of this invasive mechanical ventilation and extubation (removal of the intubation tube).

To reduce the risk of reintubation, it is recommended that a weaning test is performed prior to extubation. The purpose of this test is to simulate the conditions of breathing without the help of a ventilator after extubation. If the weaning test is successful, the patient can theoretically be extubated.

There are several causes associated with extubation failure, but studies suggest that sleep deprivation or poor sleep quality in the nights before extubation is one of them. In addition, patients with COPD often have chronic sleep disturbances or induced by their stay in the ICU (asthenia, bed rest, anxiety, sedation, etc.).

The aim of our study will be to compare the sleep characteristics of COPD patients with a failed weaning test and those with a successful test. Our hypothesis is that patients with a failed weaning test will have more sleep disturbances in the period of 72 hours before the weaning test.

DETAILED DESCRIPTION:
1. Scientific justification 1.1. Current pathological knowledge

   Chronic obstructive pulmonary disease (COPD) is a common disease that will cause more than 3 million deaths worldwide in 2019, making it the third leading cause of death worldwide. Its economic impact is significant, accounting for almost 6% of the total annual healthcare budget in the European Union.

   COPD is characterised by persistent respiratory symptoms and airflow limitation due to airway abnormalities, usually caused by significant tobacco and/or environmental exposure.

   Patients with COPD may be admitted to intensive care for acute respiratory failure due to COPD (this is a severe exacerbation of BPCO) or for reasons other than COPD.

   COPD is a common condition affecting approximately 10% of patients admitted to the ICU. The presence of COPD is an independent risk factor for increased mortality, duration of mechanical ventilation and weaning time from invasive mechanical ventilation.

   More than 25% of hospitalised patients with severe exacerbations of COPD may require admission for resuscitation. Their prognosis is poor, with 15-20% of resuscitation deaths and 20-30% of in-hospital mortality.

   Patients with COPD may require invasive mechanical ventilation during exacerbations with alveolar hypoventilation, impaired oxygenation, impaired consciousness and failure of non-invasive mechanical ventilation. Apart from exacerbations of COPD, patients may receive invasive mechanical ventilation in situations such as coma, multivisceral failure or in a perioperative context. This invasive mechanical ventilation requires the use of sedation until weaning from invasive ventilation.

   In ICU, reducing the duration of invasive mechanical ventilation is an important way of avoiding complications such as ventilator-induced lung injury, ventilator-associated pneumonia, prolonged sedation, neuromyopathy and prolonged length of stay.

   Early identification of spontaneously breathing patients may shorten extubation time and reduce the duration of mechanical ventilation. However, it is necessary to assess the risk of reintubation before extubation. In fact, extubation is a high-risk situation. Extubation failure occurs in about 10-15% of cases, but can exceed 20% in patients at high risk of extubation failure and is associated with an increase in mortality of about 30%. Patients over 65 years of age or with underlying chronic cardiac or respiratory disease are at high risk of extubation failure, and COPD is one of these common chronic respiratory diseases.

   Expert recommendations on the conditions for extubation aim to reduce the incidence of associated complications. To reduce the risk of reintubation, the recommendations suggest the systematic use of a weaning test prior to extubation. Extubation criteria combine ventilatory parameters (related to ventilator settings), respiratory, haemodynamic and neurological clinical parameters. If these criteria are met, the weaning test can be performed. The aim of this test is to reproduce as closely as possible spontaneous ventilation without assistance. If the criteria are met and the weaning test is successfully completed, the patient can theoretically be weaned.

   Weaning from invasive mechanical ventilation is a critical step in the hospitalisation of COPD patients in the ICU. And as we have previously presented, COPD is a challenging risk factor for invasive mechanical ventilation.

   In terms of weaning from invasive mechanical ventilation, recent work has improved screening for weaning difficulties in the high-risk population that is part of the COPD patient population. However, to further reduce weaning failure in COPD patients, it will be necessary to target the determinants specific to COPD patients. These determinants include chronic or acquired muscular dysfunction (particularly diaphragmatic) in the ICU, abnormalities in pre-existing ventilatory control and/or due to ICU treatments, or sleep structure abnormalities that may affect weaning in these patients.

   Regarding sleep abnormalities, quantitative and qualitative changes in sleep are common in ICU patients and normal sleep architecture may disappear. A recent study by Thille et al. suggests that the duration of invasive mechanical ventilation in patients at high risk of weaning failure should be extended from 2 to 4 days in the presence of sleep abnormalities. In addition, patients sleep quality and awakenings in the period before the weaning test are correlated with the success of the test and the success of weaning itself. A limitation of these studies is that a single sleep recording was made before or after the weaning test from invasive mechanical ventilation. This meant that sleep quality could only be analysed over a short period of time.

   COPD patients often have sleep abnormalities in the basal state, mainly due to COPD with obstructive sleep apnoea syndrome (OSAS) or nocturnal hypoventilation syndrome. Sleep deprivation or poor sleep quality may be a risk factor for failure to wean from invasive mechanical ventilation in patients with COPD. This should be investigated.

   We want to study all patients with COPD who receive invasive mechanical ventilation during resuscitation for more than 24 hours.

   1.2. Research hypotheses and expected results

   Given the previously presented data suggesting an association between changes in sleep quality and failure to wean from mechanical ventilation, our hypothesis is that failure to wean from invasive mechanical ventilation will be more frequent in COPD patients with sleep abnormalities than in those without sleep abnormalities.

   As COPD patients are frequently admitted to the ICU and are at risk of weaning failure from invasive mechanical ventilation, we wanted to specifically study this patient population.

   Our aim is to compare the sleep characteristics of COPD patients who have failed the weaning test with those who have passed the weaning test for invasive mechanical ventilation.

   Therefore, we want to record sleep and measure the presence of possible sleep abnormalities in all COPD patients receiving invasive mechanical ventilation for more than 24 hours in the intensive care unit, as soon as sedative treatments are stopped and for a period of 7 days after stopping these treatments.

   Continuous sleep recording is performed using the DREEM headband (Beacon Biosignals, Inc.), which is a practical and validated alternative to polysomnography (PSG) and allows for sleep staging with similar detail as experienced evaluators. Total sleep time and the duration of each sleep stage are measured by automated analysis of the DREEM headband. Sleep microarchitecture and the number of transitions between sleep stages are also measured by automated analysis. A weaning test for invasive mechanical ventilation is then performed according to the recommendations of the International Conference of Consensus on Weaning.

   The medical community interest in sleep quality in the ICU has increased in recent years because of the various consequences of poor sleep quality, such as ICU delirium, abnormal human ventilatory control or deregulated immune system activity. The development of new tools to assess and measure sleep quality in the ICU has been promoted in recent years, and protocols to improve sleep quality in the ICU are being developed.

   Like nutrition and pain management, improving sleep quality is an adjunctive therapy to resuscitation that should be considered in all ICU patients because of its potential impact.

   The clinical implications in this population of COPD patients at risk of complex weaning from invasive mechanical ventilation are many, and we detail the most important ones:
   * Knowing that weaned patients contribute disproportionately to ICU costs and morbidity, studies are clearly needed to determine why these abnormalities occur (sleep deprivation, metabolic factors, medications...) and how to prevent them;
   * Sleep monitoring throughout the ICU stay could allow early detection of sleep and wakefulness abnormalities so that measures can be taken to mitigate their progression;
   * Visual inspection of the electroencephalogram (EEG) does not appear to be sufficient to detect EEG abnormalities of arousal and sleep; the development of tools to assist practitioners in this detection should be encouraged;
   * Raising the awareness of ICU clinicians about the quality of sleep in ICU patients and therapeutic strategies to improve sleep, such as adapting sedation management strategies, redesigning the ICU environment and workflow, using treatments that act on circadian rhythms such as melatonin, promoting noise reduction protocols, music therapy, light therapy and the use of different mechanical ventilation methods.
2. Description of the study

   This is a human study, observational, prospective, monocentric (Medical ICU, Grenoble Alpes University Hospital).
3. Number of subjects to include

Based on a hypothesis of 70% withdrawal test failure in COPD patients with sleep abnormalities versus 30% in those without sleep abnormalities, 36 patients must be included in the study cohort to achieve 80% power with an alpha risk set at 5% in a bilateral situation. We also expected a drop-out rate of approximately 15% due to technical problems. We therefore planned to enrol 42 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with COPD according to the GOLD criteria.
* Mechanical ventilation by endotracheal tube and mechanical ventilation for > 24 hours.
* Withdrawal of treatment with continuous sedation and/or neuroleptics.
* Adequate recovery with Glasgow Coma Scale ≥ 8.

Exclusion Criteria:

* Patients with central nervous system damage or neuromuscular pathology.
* Pregnant or postpartum patients.
* Patients or their relatives who object to participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with COPD who received invasive mechanical ventilation for more than 24 hours in the intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
To identify and measure the association between the presence of abnormal sleep parameters and the outcome of weaning from invasive mechanical ventilation. | day 7
  Sleep parameters will be analysed according to a hierarchical sequential analysis with the following order
  1. No REM sleep,
  2. Atypical sleep and
  3. Sleep time.
  Results (failure or success) of the invasive mechanical ventilation test performed according to the recommendations of the International Conference on Warning Consensus.

SECONDARY OUTCOMES:
To identify for and measure the association between the presence of sleep disorders and extubation failure. | day 7
  Failure or success of extubation.
To search for and measure the association between the presence of sleep parameters and the duration of invasive mechanical ventilation after weaning from sedation. | day 7
  Duration of invasive mechanical ventilation in hours after weaning from sedation and patient awakening (Glasgow score ≥ 8).
To search for and measure the association between the presence of sleep parameters and self-extubation. | day 7
  Rate of self-extubation.
To detect and measure the association between the presence of sleep parameters and the impact of the occurrence of ventilator-acquired pneumonia after enrolment. | day 7
  Incidence of ventilator-acquired pneumonia (VAP) after enrolment.

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Marie GALERNEAU, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Grenoble Alpes University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No